CLINICAL TRIAL: NCT03887377
Title: The Efficacy and Molecular Mechanism of Botulinum Toxin in the Reduction of Breast Reduction Mammoplasty Scar Formation: A Prospective, Controlled, Randomized, Double-blinded Study
Brief Title: The Efficacy and Molecular Mechanism of Botulinum Toxin in the Reduction of Breast Reduction Mammoplasty Scar Formation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, David M. Ozog, Chair of Department of Dermatology, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 12373
Record Dates: First submitted 2019-02-20; First posted 2019-03-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Scar; Hypertrophic Scar; Mammary Disorder
Keywords: macromastia; botulinum toxin; scar prevention; scar formation
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic; Breast Diseases; Gigantomastia | interventions — Botulinum Toxins; abobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Intervention Model Description: Each patient will serve as their own control as one breast incision will be injected with botulinum toxin type A while the other will receive placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The injector, patient, and outcome assessor will be blinded to the treatment side and placebo side of injection.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Breast receiving botulinum toxin (Experimental): Following reconstruction one horizontal incisional wound will be selected to receive a series of botulinum toxin injections along the wound.
  Injection abobotulinum toxin at time of surgery, single injection time with 30 gauge needle superficially, dosage determined by length of scar 5-15U per cm
  Interventions: Drug: Botulinum Toxins
- Breast receiving placebo (Placebo Comparator): The other breast will be injected with bacteriostatic normal saline in a similar fashion to the other breast. The injector will be blinded to the contents of the syringe.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Botulinum Toxins — We will be comparing botulinum toxin following breast reduction surgery to placebo injection. We will then compare photos of each breast reduction scar at set intervals following surgery.
  Other Names: Dysport; BTXa; abobotulinumtoxinA
  Arms: Breast receiving botulinum toxin
Other: Normal saline — Normal saline will serve as the placebo control on the contralateral breast
  Other Names: Placebo
  Arms: Breast receiving placebo

SUMMARY:
1. Test the ability of botulinum toxin type A, when injected into the surgical incision at the time of surgery, to decrease postoperative scar scores compared to control (normal saline) in a double-blinded randomized control trial.
2. Investigate the mechanism of BTXa effects of scar formation by measuring micro RNA profiles at two time points in the healing process.

DETAILED DESCRIPTION:
Breast reduction mammoplasty is an increasingly popular procedure in this country due to not only the perceived cosmetic benefit of the procedure but additionally the improvement in musculoskeletal pain, headaches, sleeping difficulties, breathing, depression, self-esteem, and eating disorders. Despite these benefits, outcome satisfaction the typical inverted-T scar of the Wise pattern reduction has been limited by the resulting scar formation on the breast tissue. One study demonstrated that although 86% of patients were highly satisfied with their surgery, 65% were dissatisfied with their scars, with the majority of those dissatisfied , 65%, being bothered by the horizontal component of the scar. To address cosmetic outcomes of the procedure multiple techniques have been purposed in the literature including: superior pedicle technique, vertical mammoplasty, and circum-areolar breast reduction. By selectively injecting the horizontal component of the mammoplasty scar our analysis should be independent of surgeon surgical approach if it should include a vertical incisional scar. Aesthetic results of breast mammoplasty have also been attributed to analysis of breast meridian length, modifying areolar shape and most importantly tailoring or the medial inframammary crease. Tension across the inframammary crease requires appropriate shaping in order to reduce scar hypertrophy.

Mechanical stress from wound tension has been thought to play a major role in hypertrophic scar development. Cellular and biochemical studies have demonstrated that excessive forces on tissues are tightly linked to changes in the extracellular matrix such as the induction of wound fibrosis and inhibition of fibroblast apoptosis. Recently, botulinum toxin type A has been reported as a treatment agent to counteract these effects. Although its precise mechanism is not yet completely understood, botulinum toxin type A is thought to promote apoptosis of fibroblasts derived from hypertrophic scars, leading to reduced tensile forces. In an in vivo study, human hypertrophic scars treated with botulinum toxin type A had significantly reduced fibroblast proliferation compared to a control, and had synergistic effects with intralesional steroid injections, which is a commonly used treatment but with multiple adverse effects.

Botulinum toxin type A is a potent neurotoxin used in a wide scope of clinical settings, and has been injected for cosmetic purposes for more than two decades. Its clinical use specifically for hypertrophic scars, including those of the face, has recently been demonstrated. Furthermore, a randomized double-blinded split scar study has demonstrated the safety and efficacy of botulinum toxin type A injection into thyroidectomy scars for scar prevention. Although a well-controlled and designed study, its weaknesses include the difficult applicability of the Korean population to that of the United States, the relatively small number of patients included in the trial, the injection of botulinum toxin type A post-surgery instead of at the time of surgery (as the latter is often reported in other studies and is thought to be more beneficial). This protocol is designed to test the ability of botulinum toxin type A to improve post-surgical breast scarring in a randomized, double-blinded, controlled clinical trial at Henry Ford Hospital. It expands upon previous studies that have already demonstrated its safety and good tolerance profile, and will combine the expertise of the Dermatology department and Plastic surgeons. We will study breast reduction scars, as this will allow patients to serve as their own control group.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing breast reduction surgery
2. Does not meet any exclusion criteria
3. Female
4. >18 years old
5. Willing to participate in study

Exclusion Criteria:

1. Allergy to botulinum toxin
2. Currently pregnant or breast feeding
3. Myasthenia gravis
4. Lambert-Eaton Myasthenic Syndrome
5. Amyopathic Lateral Sclerosis
6. Previous injection of botulinum toxin in the chest area within 6 months prior to enrollment
7. History of keloid or hypertrophic scar
8. History of previous breast surgery with scar affecting inframammary skin
9. Male Sex
10. Refusal to participate in the study
11. Unable to make follow up appointments up to 6 months
12. Less than 18 years of age
13. History of radiation to the breast

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Modified Patient and Observer Scar Assessment Scale v2.0 (POSAS) | Photos will be reviewed at the 1 week follow surgery
  Two blinded dermatologists will make the objective clinical assessments separately using a modified POSAS Patient and Observer Scar Assessment Scale v2.0
  It includes assessing the vascularity, pigmentation, thickness, relief, and surface area from a scale from 1 to 10. Pliability, which is included in the original scale, will be excluded for this study given the use of photographs for assessment. The scale also includes the patient's opinion of their own scar, which includes pain, pruritis, color, stiffness, thickness, irregularity from a scale from 1 to 10.Independent objective review of scar photos will be graded on a scale 1-10. 1 is normal skin. 10 is worst scar imaginable.
Modified Patient and Observer Scar Assessment Scale v2.0 (POSAS) | 4-8 weeks following surgery
  Two blinded dermatologists will make the objective clinical assessments separately using a modified POSAS Patient and Observer Scar Assessment Scale v2.0
  It includes assessing the vascularity, pigmentation, thickness, relief, and surface area from a scale from 1 to 10. Pliability, which is included in the original scale, will be excluded for this study given the use of photographs for assessment. The scale also includes the patient's opinion of their own scar, which includes pain, pruritis, color, stiffness, thickness, irregularity from a scale from 1 to 10.Independent objective review of scar photos will be graded on a scale 1-10. 1 is normal skin. 10 is worst scar imaginable.
  These scores will be compared to the 1 week time point.
Modified Patient and Observer Scar Assessment Scale v2.0 (POSAS) | 6 month mark following surgery
  Two blinded dermatologists will make the objective clinical assessments separately using a modified POSAS Patient and Observer Scar Assessment Scale v2.0
  It includes assessing the vascularity, pigmentation, thickness, relief, and surface area from a scale from 1 to 10. Pliability, which is included in the original scale, will be excluded for this study given the use of photographs for assessment. The scale also includes the patient's opinion of their own scar, which includes pain, pruritis, color, stiffness, thickness, irregularity from a scale from 1 to 10.Independent objective review of scar photos will be graded on a scale 1-10. 1 is normal skin. 10 is worst scar imaginable.
  These scores will be compared to the 1 week and the 4-8 weeks time point.

CONTACTS AND LOCATIONS:
Overall Officials: David Ozog, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There will be a publication based on the results of the study. We will not be sharing individual participant data outside of our facility. All data will be kept on the secure drive at Henry Ford Health Systems.

REFERENCES:
- [Result] Singh KA, Losken A. Additional benefits of reduction mammaplasty: a systematic review of the literature. Plast Reconstr Surg. 2012 Mar;129(3):562-570. doi: 10.1097/PRS.0b013e31824129ee. PMID 22090252
- [Result] Sprole AM, Adepoju I, Ascherman J, Gayle LB, Grant RT, Talmor M. Horizontal or vertical? an evaluation of patient preferences for reduction mammaplasty scars. Aesthet Surg J. 2007 May-Jun;27(3):257-62. doi: 10.1016/j.asj.2007.04.007. PMID 19341651
- [Result] Saleem L, John JR. Unfavourable results following reduction mammoplasty. Indian J Plast Surg. 2013 May;46(2):401-7. doi: 10.4103/0970-0358.118620. PMID 24501476
- [Result] Hidalgo DA. Improving safety and aesthetic results in inverted T scar breast reduction. Plast Reconstr Surg. 1999 Mar;103(3):874-86; discussion 887-9. PMID 10077078
- [Result] Wolfram D, Tzankov A, Pulzl P, Piza-Katzer H. Hypertrophic scars and keloids--a review of their pathophysiology, risk factors, and therapeutic management. Dermatol Surg. 2009 Feb;35(2):171-81. doi: 10.1111/j.1524-4725.2008.34406.x. PMID 19215252
- [Result] Niland S, Cremer A, Fluck J, Eble JA, Krieg T, Sollberg S. Contraction-dependent apoptosis of normal dermal fibroblasts. J Invest Dermatol. 2001 May;116(5):686-92. doi: 10.1046/j.1523-1747.2001.01342.x. PMID 11348456
- [Result] Chen CS. Mechanotransduction - a field pulling together? J Cell Sci. 2008 Oct 15;121(Pt 20):3285-92. doi: 10.1242/jcs.023507. PMID 18843115
- [Result] Gabbiani G. The myofibroblast in wound healing and fibrocontractive diseases. J Pathol. 2003 Jul;200(4):500-3. doi: 10.1002/path.1427. PMID 12845617
- [Result] Zhibo X, Miaobo Z. Botulinum toxin type A affects cell cycle distribution of fibroblasts derived from hypertrophic scar. J Plast Reconstr Aesthet Surg. 2008 Sep;61(9):1128-9. doi: 10.1016/j.bjps.2008.05.003. Epub 2008 Jun 13. No abstract available. PMID 18555763
- [Result] Zhibo X, Miaobo Z. Potential therapeutical effects of botulinum toxin type A in keloid management. Med Hypotheses. 2008 Oct;71(4):623. doi: 10.1016/j.mehy.2008.04.018. Epub 2008 Jun 4. No abstract available. PMID 18534768
- [Result] Xiao Z, Zhang F, Lin W, Zhang M, Liu Y. Effect of botulinum toxin type A on transforming growth factor beta1 in fibroblasts derived from hypertrophic scar: a preliminary report. Aesthetic Plast Surg. 2010 Aug;34(4):424-7. doi: 10.1007/s00266-009-9423-z. Epub 2009 Oct 3. PMID 19802513
- [Result] Chen HC, Yen CI, Yang SY, Chang CJ, Yang JY, Chang SY, Chuang SS, Hsiao YC. Comparison of Steroid and Botulinum Toxin Type A Monotherapy with Combination Therapy for Treating Human Hypertrophic Scars in an Animal Model. Plast Reconstr Surg. 2017 Jul;140(1):43e-49e. doi: 10.1097/PRS.0000000000003426. PMID 28654594
- [Result] Feily A, Fallahi H, Zandian D, Kalantar H. A succinct review of botulinum toxin in dermatology; update of cosmetic and noncosmetic use. J Cosmet Dermatol. 2011 Mar;10(1):58-67. doi: 10.1111/j.1473-2165.2010.00545.x. PMID 21332916
- [Result] Jablonka EM, Sherris DA, Gassner HG. Botulinum toxin to minimize facial scarring. Facial Plast Surg. 2012 Oct;28(5):525-35. doi: 10.1055/s-0032-1325641. Epub 2012 Oct 1. PMID 23027220
- [Result] Liu RK, Li CH, Zou SJ. Reducing scar formation after lip repair by injecting botulinum toxin. Plast Reconstr Surg. 2010 May;125(5):1573-1574. doi: 10.1097/PRS.0b013e3181d51404. No abstract available. PMID 20440184
- [Result] Zhibo X, Miaobo Z. Intralesional botulinum toxin type A injection as a new treatment measure for keloids. Plast Reconstr Surg. 2009 Nov;124(5):275e-277e. doi: 10.1097/PRS.0b013e3181b98ee7. No abstract available. PMID 20009818
- [Result] Kim YS, Lee HJ, Cho SH, Lee JD, Kim HS. Early postoperative treatment of thyroidectomy scars using botulinum toxin: a split-scar, double-blind randomized controlled trial. Wound Repair Regen. 2014 Sep-Oct;22(5):605-12. doi: 10.1111/wrr.12204. Epub 2014 Aug 26. PMID 24898579
- [Result] Larrabee WF Jr. Treatment of Facial Wounds with Botulinum Toxin A Improves Cosmetic Outcome in Primates. Plast Reconstr Surg. 2000 May;105(6):1954-1955. doi: 10.1097/00006534-200005000-00006. No abstract available. PMID 11242330
- [Result] Ziade M, Domergue S, Batifol D, Jreige R, Sebbane M, Goudot P, Yachouh J. Use of botulinum toxin type A to improve treatment of facial wounds: a prospective randomised study. J Plast Reconstr Aesthet Surg. 2013 Feb;66(2):209-14. doi: 10.1016/j.bjps.2012.09.012. Epub 2012 Oct 25. PMID 23102873
- [Result] Austin E, Koo E, Jagdeo J. The Cellular Response of Keloids and Hypertrophic Scars to Botulinum Toxin A: A Comprehensive Literature Review. Dermatol Surg. 2018 Feb;44(2):149-157. doi: 10.1097/DSS.0000000000001360. PMID 29401161
- [Result] Qu L, Liu A, Zhou L, He C, Grossman PH, Moy RL, Mi QS, Ozog D. Clinical and molecular effects on mature burn scars after treatment with a fractional CO(2) laser. Lasers Surg Med. 2012 Sep;44(7):517-24. doi: 10.1002/lsm.22055. Epub 2012 Jul 31. PMID 22907286